CLINICAL TRIAL: NCT03624699
Title: A Prospective, Unmasked, Single-Site Investigation of the iStent Inject® Devices Implanted in Combination With Cataract Surgery in Patients With Open-Angle Glaucoma
Brief Title: Investigation of the iStent Inject® Devices in Open-Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kaweh Mansouri (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor-Investigator, Dr. Kaweh Mansouri, Sponsor-Investigator, Primary investigator, Swiss Vision Network
Organization: Swiss Vision Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLK-iStent-inject
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma, Open-Angle
Keywords: glaucoma; Minimally Invasive Glaucoma Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: Historic control (before vs. after intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Glaukos iStent inject® (Experimental): Patients suffering from cataract and open-angle glaucoma. Glaukos iStent inject® is implanted during routine cataract surgery. The effect on IOP/glaucoma medications is monitored.
  Interventions: Device: Glaukos iStent inject®

INTERVENTIONS:
Device: Glaukos iStent inject® — iStent inject® Devices Implanted in Combination with Cataract Surgery in Patients with Open-Angle Glaucoma

SUMMARY:
The aim of this study is to evaluate the safety and intraocular pressure (IOP) lowering effect of two iStent inject devices in combination with cataract surgery in patients with mild-to-moderate open-angle glaucoma.

DETAILED DESCRIPTION:
Patients suffering from open-angle glaucoma who are planning to undergo cataract surgery and are matching the inclusion criteria will be offered to join the study until the desired sample size (50) is reached. Combined cataract-iStent surgery will be performed as per the devices' manufacturers' instructions. Two iStent inject devices will be micro-invasively implanted in the trabecular meshwork of the eye during planned cataract surgery. Six post-operative follow-ups will be carried out over a duration of 12 months, during which various measurements will be made. Performance Outcomes will analyse the proportion of patients with IOP reduction of ≥ 20% vs. baseline mean IOP, at 6 and 12 months. Quality of life outcome will look at the improvement in perceived quality of life as expressed in the NEI VFQ-25 questionnaires from baseline to 3 and 12 months. The rate of adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma, pseudoexfoliative glaucoma, or pigmentary glaucoma
* Mild to moderate glaucoma (defined as C/D ratio ≤ 0.8)
* Phakic eye requiring cataract surgery
* Preoperative IOP up to 30 mmHg (medicated or not)
* Patients with side-effects to, or complications from, medications
* Patients who would benefit from a reduction of IOP and/or reduction of medication
* Normal angle anatomy as determined by gonioscopy;
* Absence of peripheral anterior synechiae (PAS), rubeosis or other angle abnormalities that could impair proper placement of iStent inject device
* Able and willing to attend scheduled follow-up exams for 12 months postoperatively
* Able and willing to provide written informed consent on the approved Informed Consent Form

Exclusion Criteria:

* Inclusion of the fellow eye in this study (only one eye per subject)
* Aphakic patients or pseudophakic patients
* Prior stent implantations in the study eye
* Eyes with primary angle closure glaucoma, or any secondary angle closure glaucoma
* Traumatic or uveitic glaucoma; or any glaucoma associated with vascular disorders
* Patients with any type of condition that may cause elevated episcleral venous pressure
* Functionally significant visual field loss, including severe nerve fiber bundle defects such as Bjerrum scotoma
* Prior glaucoma treatment (laser or surgery)
* Any active corneal inflammation, edema, or opacity severe-enough to impair gonioscopy / fundus examination
* Any pathology for which, in the investigator's judgment, the following would be either at risk or contraindicated:

  * stent implantation,
  * compliance to elements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Performance Outcome: IOP reduction | 12 months
  Proportion of patients with IOP reduction of ≥ 20% vs. baseline mean IOP, at 12 months.

SECONDARY OUTCOMES:
Quality of life: NEI VFQ-25 score | 12 months
  Improvement in perceived quality of life as expressed in the NEI VFQ-25 (National Eye Institute Vision Function) questionnaires from baseline to 12 months.
Safety Outcome: Adverse events | 12 months
  Rate of adverse events through the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, MD MPH, Study Director — Glaucoma Research Centre, Montchoisi Clinic, Lausanne; André Mermoud, MD, Study Director — Glaucoma Research Centre, Montchoisi Clinic, Lausanne
Locations (1):
- Glaucoma Research Centre, Montchoisi Clinic, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillmann K, Mansouri K, Ambresin A, Bravetti GE, Mermoud A. A Prospective Analysis of iStent Inject Microstent Implantation: Surgical Outcomes, Endothelial Cell Density, and Device Position at 12 Months. J Glaucoma. 2020 Aug;29(8):639-647. doi: 10.1097/IJG.0000000000001546. PMID 32433094